CLINICAL TRIAL: NCT05312996
Title: Perceived Stress and Patterns of Autonomic Function: a Protocol Development Study
Brief Title: Autonomic Nervous System Function - Hypertension
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Prioritizing other studies
Sponsor: Life University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: I-0017
Record Dates: First submitted 2022-03-02; First posted 2022-04-06 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Galvanic Skin Response

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypertension (Experimental): Hypertension test group.
  Interventions: Other: Heart Rate Variability; Other: Galvanic Skin Response (Biopac)
- Active Comparator (Other): Non Hypertension compare group.
  Interventions: Other: Heart Rate Variability; Other: Galvanic Skin Response (Biopac)

INTERVENTIONS:
Other: Heart Rate Variability — Caretaker Heart Rate Variability ECG wrist monitor and chest patch.
Other: Galvanic Skin Response (Biopac) — Galvanic Skin Response- measuring autonomic response-via perspiration

SUMMARY:
The Life University Center for Chiropractic Research is conducting a research study to better understand the physiological differences, in terms of Autonomic nervous system function, between individuals with Hypertension and control individuals with out hypertension. Data will be gathered using Heart Rate Variability (HRV), and Galvanic Skin Response (GSR). A series of tests will be conducted to elicit Autonomic Nervous system responses. These tests include Cold Face Test (mammalian dive reflex), Cold Pressor test, Sit to stand, and the Valsalva maneuver.

DETAILED DESCRIPTION:
The objective of the study is to ascertain the level of autonomic health in persons with hypertension versus a healthy population. Further, via the implemented protocol, the study will attempt to develop a sequence of autonomic nervous system tests to be used in future studies and clinical settings

ELIGIBILITY:
Participants will be included in the hypertension group if they present with the following:

* Hypertension, defined as:
* Self-reported or previously diagnosed with elevated resting state blood pressure (120-129 systolic and less than 80 mmHg diastolic) or stage 1 hypertension with a blood pressure of Systolic between 130- and 139-mm Hg with a diastolic of 80-89 mmHg.
* Or medically diagnosed and managed stage 2 hypertension with blood pressure of Systolic between 140- and 159-mm Hg or diastolic 90 and 99 mm
* between the ages of 18-65
* Able to wear a monitor on their right wrist.
* Able to wear a pulse oximeter on their left hand.

Participants will be included in the healthy group if they present with the following:

* between the ages of 18-65
* Able to wear a monitor on their right wrist.
* Able to wear a pulse oximeter on their left hand.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-10-26 (Estimated); Study Completion 2023-10-26 (Estimated)

PRIMARY OUTCOMES:
Heart Rate Varability | Through study completion, an average of 1 year
  Caretaker Heart Rate Variability (HRV) Electrocardiogram (ECG) wrist monitor and chest patch.
Galvanic Skin Response | Through study completion, an average of 1 year
  Galvanic Skin Response- measuring autonomic response-via perspiration

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Sullivan, DC, PhD, Study Director — Life Univeristy
Locations (1):
- Dr. Sid E. Williams Center for Chiropractic Research, Atlanta, Georgia, United States